CLINICAL TRIAL: NCT02373475
Title: Effect of Perioperative Lung Protective Strategies on the Occurrence of Postoperative Pulmonary Complications in Patients Undergoing Lumbar Spinal Surgery in the Prone Position
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2014-0955
Record Dates: First submitted 2015-02-10; First posted 2015-02-27 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Complications
Keywords: spine surgery; prone position; intraoperative lung protective strategies; postoperative pulmonary complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional ventilation (Experimental): Conventional ventilation with TV of 10 mL/kg predicted body weight (PBW) without positive end-expiratory pressure (PEEP) during the surgery under general anesthesia
  Interventions: Other: Conventional ventilation
- Protective lung ventilation (Active Comparator): Protective lung ventilation with TV of 6 mL/kg PBW, PEEP of 6 cmH2O and recruitment maneuver during the surgery under general anesthesia
  Interventions: Other: Protective lung ventilation

INTERVENTIONS:
Other: Conventional ventilation — Conventional ventilation with TV of 10 mL/kg predicted body weight (PBW) without positive end-expiratory pressure (PEEP) during the surgery under general anesthesia
  Arms: Conventional ventilation
Other: Protective lung ventilation — Protective lung ventilation with TV of 6 mL/kg PBW, PEEP of 6 cmH2O and recruitment maneuver during the surgery under general anesthesia
  Arms: Protective lung ventilation

SUMMARY:
Postoperative pulmonary complications are main cause of overall perioperative morbidity and mortality in the patients following general anesthesia. A protective ventilation strategy refers to the use of low VT (in the range of 4-8 ml/kg of the predicted body weight) with positive end-expiratory pressure (PEEP), with or without recruitment maneuver. Protective ventilation has been considered the optimal practice in patients suffering from the acute respiratory distress syndrome (ARDS). However, few human studies have assessed how to ventilate healthy lungs in patients undergoing general anesthesia, especially in prone position. Prior studies reported that in the patients undergoing major abdominal surgery in supine position, intraoperative lung protective ventilator settings had the potential to protect against pulmonary complications. Therefore, the investigators planned this study to better specify the effect of intraoperative protective ventilation in surgical patients in the prone position.

ELIGIBILITY:
Inclusion Criteria:

* the patient undergoing elective lumbar spine surgery of two hours or more in the prone position
* the age: 19 yrs and older
* the patients had a preoperative risk index for pulmonary complications of more than 2.

Exclusion Criteria:

* Patients with altered mental status or increased intracranial pressure
* Body mass index more than 35 kg/m2
* Patients with persistent hemodynamic instability or intractable shock
* Severe cardiac disease defined as New York Heart Association class III or IV or acute coronary syndrome or persistent ventricular tachyarrhythmias
* Recent history of invasive ventilation (within two weeks)
* Recent history of pneumonia, ALI/ARDS or sepsis (within two weeks)
* History of pulmonary resection, emphysema or chronic obstructive pulmonary disease (COPD)
* Repeated systemic corticosteroid therapy for acute exacerbations of COPD or asthma
* Recent immunosuppressive medication defined as need of chemotherapy or radiation therapy (within two months)
* History of neuromuscular disease
* Emergency operation
* Patient refusal
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
forced vital capacity (FVC) | 3 days after the spine surgery
  The changes in the pulmonary functional tests [forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1)].Pulmonary functional tests were performed at the bedside by using a spirometer while the patients in a seated, comfortable position.
forced expiratory volume in 1 second (FEV1) | 3 days after the spine surgery
  The changes in the pulmonary functional tests [forced vital capacity (FVC) and forced expiratory volume in 1 second (FEV1)].Pulmonary functional tests were performed at the bedside by using a spirometer while the patients in a seated, comfortable position.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea